CLINICAL TRIAL: NCT00290368
Title: Assessment of Inflammatory Mediator and Cellular Changes Following Repeated Nasal Allergen Challenge in Subjects With Allergic Rhinitis Sensitive to Timothy Grass Pollen - a Validation Study
Brief Title: Repeat Nasal Allergen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CPJMR0052104
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Hayfever
Keywords: Nasal allergen challenge; Allergic rhinitis; Timothy grass pollen; inflammatory mediators
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Patch Tests; Nasal Lavage

INTERVENTIONS:
Procedure: Skin Prick Test
Procedure: Nasal allergen challenge
Procedure: Nasal filter paper placement
Procedure: Nasal lavage
Procedure: Nasal scrape
Procedure: Nasal symptoms score

SUMMARY:
This is a non-drug, biomarker study to assess the utility of the model of repeated nasal allergen challenges in subjects with atopic rhinitis as a method of inducing an increased response to inhaled allergen, which will more closely resemble the responses seen during the hayfever season.

DETAILED DESCRIPTION:
This is a non-drug, biomarker study to assess the utility of the model of repeated nasal allergen challenges in subjects with atopic rhinitis as a method of inducing an increased response to inhaled allergen, which will more closely resemble the responses seen during the hayfever season.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with a history of seasonal (intermittent) atopic rhinitis, aged 18-40 years.
2. Otherwise healthy with no health problems that may jeopardize the subjects participating in the study, absence of history of other significant allergies.

Exclusion Criteria:

1. Smokers (use of tobacco products in the previous 3 months).
2. Presence of any respiratory disease other than a history of mild stable asthma not requiring treatment and associated with normal lung function (FEV1 > 80% predicted at screening).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2006-02; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: Trevor T Hansel, FRCPath, Principal Investigator — Imperial College London
Locations (1):
- National Heart & Lung Institute Clinical Studies Unit, London, United Kingdom